CLINICAL TRIAL: NCT05535205
Title: Effectiveness and Costs of a Digital Versus Face-to-face Preoperative Assessment Clinic: a Non-inferiority Trial
Brief Title: Effectiveness and Costs of a Digital Versus Face-to-face Preoperative Assessment Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonessenhuis, Utrecht (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 21-010
Record Dates: First submitted 2022-09-05; First posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Surgery
Keywords: Preoperative assessment clinic; Preoperative anesthetic screening; Patients requiring surgery; Surgical patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Face-to-face preoperative assessment group (Active Comparator): The face-to-face screening consist of two 20-minute consecutive consultations with a nurse and subsequently an anesthesiologist or PA. The nurse obtains basic patient health information, provides information on the upcoming hospital admission, and gives advice in lifestyle procedures around the surgery. The physician assesses the patient's health status based on co-morbidities, medication use, previous surgery, and lifestyle habits to predict preoperative risks and determine the optimal anesthetic technique. Additional diagnostics, such as blood tests or electrocardiogram, can be ordered and optional anesthetic techniques will subsequently be presented and discussed with the patient, after which informed consent will be obtained.
  Interventions: Other: Face-to-face preoperative assessment
- Digital preoperative assessment group (Active Comparator): Patients in the digital preoperative assessment group are asked to complete an electronic screening questionnaire through the digital patient portal of the hospital. The questionnaire was designed by the anesthetic department physicians and consisted of 50 health related questions. Through the same digital patient portal, patients have access to animated instructional videos that provides information on anesthetic techniques, preoperative lifestyle advises and procedures around the upcoming surgery. The videos can be reviewed at any desired moment in time. A telephone appointment is scheduled solemnly to decide on the anesthesia technique and obtain informed consent since this process was technically not available in the electronic portal. Physicians were thoroughly instructed not to provide more information or answer questions. Patients are instructed to complete the electronic screening questionnaire and assess the animated videos before the scheduled appointment with the physician.
  Interventions: Other: Digital preoperative assessment

INTERVENTIONS:
Other: Digital preoperative assessment — a digital preoperative assessment for patient requiring surgery
  Arms: Digital preoperative assessment group
Other: Face-to-face preoperative assessment — a face-to-face preoperative assessment for patient requiring surgery
  Arms: Face-to-face preoperative assessment group

SUMMARY:
A digital preoperative assessment clinic provides a solution for the increasing demand and declining performance on waiting times for surgery, while conducting assessments to a high standard. However, it remains unclear if a digital preoperative assessment is as effective as a face-to-face clinic in terms of patient health outcomes and experience compared. This study aimed to compare quality or recovery and overall patient experience in patients undergoing a digital preoperative assessment versus regular face-to-face consultations.

DETAILED DESCRIPTION:
Study design This is a randomized (1:1), open label, noninferiority trial performed at 2 locations of a Dutch, urban, secondary care hospital.

Aims

1. demonstrate the noninferiority of a digital PAC, in terms of postoperative quality of recovery, compared with a face-to-face PAC, and
2. demonstrate if there is a difference in preoperative anxiety, decisional conflict, patient satisfaction, morbidity, mortality, American Society of Anesthesiologists score (ASA) reliability, and costs.

Study population Participants aged 18 and older admitted to the PAC department with a request of undergoing surgery were evaluated for study enrollment. The trial inclusion criteria are age 18 and older, ASA classification I to IV, fluent in Dutch, the availability of an online personal computer at home, and able to give informed consent. Exclusion criteria are pregnant women, and patients undergoing a non-standard pre-operative assessment procedure which included breast- and gastrointestinal oncology and cardiac procedures.

Outcomes Primary: Quality of recovery 40 (QOR-40) scale assessed at 48 hours postoperative.

Secondary outcomes (Measured 1 day prior to surgery):

* State-Trait Anxiety Inventory (STAI) form Y1 (also at baseline)
* Decisional conflict scale (DCS)
* Patient satisfaction with information (NR 1-10)
* Patient satisfaction with the screening process (NR 1-10) Measured during the study
* ASA reliability
* Postoperative length of stay
* 30-day complications
* 30-day mortality
* preoperative anesthetic assessment and surgery cancelation
* loan costs

Sample size This sample size calculation will be based on noninferiority tests for the continuous primary outcome quality of recovery score (QoR-40) measured at 48 hours after surgery. The noninferiority margin is set at -6 points, which is based on a study by Myles et al. who found a minimal clinical important difference (MCID) of 6.3 for the QOR-40 questionnaire, which was subsequently rounded down. Based on this study, the expected QoR-40 score was177 with a standard deviation of 16 on postoperative day 2 for the control group (face-to-face consultations). A total of 224 patients, 112 in each group, would yield a power of 80%, using a one-sided 97,5% confidence interval (CI), to establish whether a digital PAC is noninferior compared to a face-to-face PAC. With an estimated dropout rate of 25%, a total of 299 patients (150 patients per group) need to be enrolled.

Analysis Data will be analyzed as per-protocol. A linear mixed effects model will be conducted with study group and QOR-baseline as fixed effects and treating specialism as random effect. The primary outcome of QoR-40 will be presented as the mean difference between study groups (digital screening - face-to-face screening) with the upper and lower bound of the 95% CI and will be labelled non-inferior when the non-inferiority margin of -6 lies outside the lower bound of the 95% CI. CIs will be calculated using linear regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* patients to the PAC department with a request of undergoing surgery
* 18 and older
* ASA classification I to IV
* general surgery (vascular, traumatic, gastrointestinal, oncological), gynecology, otolaryngology, neurosurgery, plastic surgery, orthopedics, and ophthalmology.
* fluent in Dutch
* the availability of an online personal computer at home
* and able to give informed consent.

Exclusion Criteria:

* pregnant women
* patients undergoing a non-standard pre-operative assessment procedure which included breast- and gastrointestinal oncology and cardiac procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Quality of recovery 40 (QOR-40) scale | Measured 48 hours postoperative
  The QoR-40 is a validated composite endpoint that can be used to evaluate anesthetic or surgical procedure. The questionnaire consists of 40 questions on a 5-point Likert scale that provides a global score and sub scores across five dimensions: patient support, comfort, emotions, physical independence, and pain. The highest achievable score, indicating maximum quality of recovery, is 200. The lowest score, indicating worst quality of recovery, is 40. The questions are related to the quality of recovery over the past 24 hours.

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory (STAI) form Y1 | Measured at 24 hours preoperative
  A psychological inventory consisting of 40 self-report items on a 4-point Likert scale. The STAI measures two types of anxiety - state anxiety and trait anxiety. Higher scores are positively correlated with higher levels of anxiety. The range of possible scores of the STAI varies from a minimum score of 20 (minimum anxiety) to a maximum score of 80 (maximum anxiety)
Decisional conflict scale (DCS) | Measured at 24 hours preoperative
  The decisional conflict scale (DCS) measures personal perceptions of:
  uncertainty in choosing options; modifiable factors contributing to uncertainty such as feeling uninformed, unclear about personal values and unsupported in decision making; and effective decision making (in full version) such as feeling the choice is informed, values-based, likely to be implemented and expressing satisfaction with the choice.
  Scores range from 0, no decisional conflict, to 100, extremely high decisional conflict.
Patient satisfaction with the information | Measured at 24 hours preoperative
  On a NR-scale from 1-10. 1 is least satisfied, 10 is most satisfied.
Patient satisfaction with the entire screening process | Measured at 24 hours preoperative
  On a NR-scale from 1-10. 1 is least satisfied, 10 is most satisfied.
ASA score reliability | During the PAC and just before surgery (1-2 hours)
  Reliability of the ASA score administered by the physician during the PAC and the ASA score administered by the physician just before surgery. Reliability is presented as quadratic weighted kappa values: 0 is low agreement, 1 is perfect agreement.
Postoperative length of stay | until 30 days after surgery
  in days
30-day complications and mortality | until 30 days after surgery
  Complications due to surgery or anesthesia are registered, as well as 30-day mortality
Cancelation of PAC appointment or cancelation of surgery | This is measured from moment of randomization to moment of surgery, which is on average 2 months from randomization.
  Number of PAC appointment cancellations and cancelled surgeries. Each cancelled appointment of surgery is registered in the medical record an retrospectively assessed.
Loan costs | until 30 days after surgery
  Difference in loan costs of nurses and physicians

CONTACTS AND LOCATIONS:
Overall Officials: Reinier Tromp Meesters, Msc, Study Chair — Diakonessenhuis, Utrecht; Mark van Heijl, PhD, Study Chair — Diakonessenhuis, Utrecht
Locations (1):
- Diakonessenhuis, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van den Blink A, Janssen LMJ, Hermanides J, Loer SA, Straat FK, Jessurun EN, Schwarte LA, Schober P. Evaluation of electronic screening in the preoperative process. J Clin Anesth. 2022 Nov;82:110941. doi: 10.1016/j.jclinane.2022.110941. Epub 2022 Aug 5. PMID 35939972
- [Result] Milne-Ives M, Leyden J, Maramba I, Chatterjee A, Meinert E. The Potential Impacts of a Digital Preoperative Assessment Service on Appointments, Travel-Related Carbon Dioxide Emissions, and User Experience: Case Study. JMIR Perioper Med. 2022 Feb 16;5(1):e28612. doi: 10.2196/28612. PMID 35171104
- [Result] Blanco Vargas D, Faura Messa A, Izquierdo Tugas E, Santa-Olalla Bergua M, Noguera Sopena MM, Manoso Noriego M. [Online versus non-standard face to face preoperative assessment: cost effectiveness]. Rev Esp Anestesiol Reanim. 2012 Aug-Sep;59(7):350-6. doi: 10.1016/j.redar.2012.05.039. Epub 2012 Jul 10. Spanish. PMID 22784647
- [Result] Howell M, Hood AJ, Jayne DG. Use of a patient completed iPad questionnaire to improve pre-operative assessment. J Clin Monit Comput. 2017 Feb;31(1):221-225. doi: 10.1007/s10877-015-9818-0. Epub 2015 Dec 29. PMID 26715416
- [Result] Taylor SK, Andrzejowski JC, Wiles MD, Bland S, Jones GL, Radley SC. A prospective observational study of the impact of an electronic questionnaire (ePAQ-PO) on the duration of nurse-led pre-operative assessment and patient satisfaction. PLoS One. 2018 Oct 19;13(10):e0205439. doi: 10.1371/journal.pone.0205439. eCollection 2018. PMID 30339687
- [Result] Osman T, Lew E, Lum EP, van Galen L, Dabas R, Sng BL, Car J. PreAnaesThesia computerized health (PATCH) assessment: development and validation. BMC Anesthesiol. 2020 Nov 14;20(1):286. doi: 10.1186/s12871-020-01202-8. PMID 33189131
- [Derived] van Hoorn BT, Tromp DJ, van Rees RCM, van Rossenberg LX, Cazemier HK, van Heijl M, Tromp Meesters RC. Effectiveness of a digital vs face-to-face preoperative assessment: A randomized, noninferiority clinical trial. J Clin Anesth. 2023 Nov;90:111192. doi: 10.1016/j.jclinane.2023.111192. Epub 2023 Jul 18. PMID 37467628